CLINICAL TRIAL: NCT00229073
Title: A Placebo-Controlled, Double-Blind, Randomized, Parallel-Group Study Of The Efficacy And Safety Of Dapoxetine In The Treatment Of Subjects With Premature Ejaculation
Brief Title: A Study of the Effectiveness and Safety of Dapoxetine in the Treatment of Men With Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004231
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Erectile Dysfunction
Keywords: dapoxetine; premature ejaculation; ejaculation; sexual dysfunction; orgasmic disorder; sexual intercourse
MeSH Terms: conditions — Erectile Dysfunction; Premature Ejaculation; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Coitus | interventions — dapoxetine

INTERVENTIONS:
Drug: dapoxetine

SUMMARY:
The primary purpose of the study is to demonstrate that dapoxetine can prolong intravaginal ejaculatory latency time (IELT) compared with placebo in men with premature ejaculation (PE).

DETAILED DESCRIPTION:
Premature ejaculation (PE) is a form of male sexual dysfunction. An objective measurement of PE in clinical studies is the intravaginal ejaculatory latency time (IELT). This is a multicenter, placebo-controlled, double-blind, randomized, parallel-group study in men with PE. The study will consist 3 phases: pre-randomization phase (a screening visit and a 4-week baseline period); 24-week double-blind treatment phase during which patients will receive dapoxetine or placebo for use on an "as-needed" basis; and, 1-week double-blind withdrawal phase (dapoxetine or placebo) with a post-study telephone contact approximately 2 weeks after the end of treatment. The total duration of the study is approximately 31 weeks. Assessments of effectiveness include the average intravaginal ejaculatory latency time, as measured by stopwatch during sexual intercourse, during the treatment period; control over ejaculation, satisfaction with sexual intercourse, and severity of symptoms, based on questions asked at monthly intervals through the treatment phase. Safety assessments include the incidence, severity, and type of adverse events throughout treatment and follow up (Week 27), as well as laboratory tests and questionnaires to monitor possible changes in mood, anxiety, motor responses, and sexual function at specified times during the study. The study hypothesis is that treatment for 24 weeks with dapoxetine prolongs intravaginal ejaculatory latency time, compared with placebo, in men with PE. Oral tablets of dapoxetine (30 milligrams[mg] or 60mg) or placebo taken as needed during 24 weeks of treatment. No more than 1 dose within a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in a stable, monogamous sexual relationship with the same woman for at least 6 months and plans to maintain this relationship for the duration of the study
* diagnosis of premature ejaculation (PE) according to the criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) for at least 6 months before study initiation
* history of intravaginal ejaculatory latency time (IELT) of <2 minutes in at least 3 out of 4 events
* good general health
* patient's partner must have a negative urine pregnancy test at time of screening

Exclusion Criteria:

* Not taken dapoxetine or participated in another study investigating pharmacologic treatment of PE within the last 3 months
* no history of any medical events that are associated with the development of PE
* not taken another investigational drug within 1 month, or used an experimental medical device within 6 months, of study initiation
* no positive diagnosis of depressive or anxiety disorder, manic episode, panic disorder, obsessive-compulsive disorder, posttraumatic stress disorder, alcohol abuse and dependence, schizophrenia, or other psychotic disorders
* no known allergy or hypersensitivity to selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2004-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Average Intravaginal ejaculatory latency time (IELT), as measured by stopwatch, during sexual intercourse, at the end of the treatment period (week 24)

SECONDARY OUTCOMES:
Control over ejaculation, satisfaction with sexual intercourse, and severity of symptom impressions, based on questions asked at monthly intervals through Week 24; incidence, severity, and type of adverse events throughout study and follow up (Week 27)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Buvat J, Tesfaye F, Rothman M, Rivas DA, Giuliano F. Dapoxetine for the treatment of premature ejaculation: results from a randomized, double-blind, placebo-controlled phase 3 trial in 22 countries. Eur Urol. 2009 Apr;55(4):957-67. doi: 10.1016/j.eururo.2009.01.025. Epub 2009 Jan 21. PMID 19195772
- [Derived] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176
- [Derived] Porst H, McMahon CG, Althof SE, Sharlip I, Bull S, Aquilina JW, Tesfaye F, Rivas DA. Baseline characteristics and treatment outcomes for men with acquired or lifelong premature ejaculation with mild or no erectile dysfunction: integrated analyses of two phase 3 dapoxetine trials. J Sex Med. 2010 Jun;7(6):2231-2242. doi: 10.1111/j.1743-6109.2010.01820.x. Epub 2010 Apr 19. PMID 20412423
- [Derived] Althof SE, Brock GB, Rosen RC, Rowland DL, Aquilina JW, Rothman M, Tesfaye F, Bull S. Validity of the patient-reported Clinical Global Impression of Change as a measure of treatment response in men with premature ejaculation. J Sex Med. 2010 Jun;7(6):2243-2252. doi: 10.1111/j.1743-6109.2010.01793.x. Epub 2010 Mar 30. PMID 20367770
- See also: A Placebo-Controlled, Double-Blind, Randomized, Parallel-Group Study of the Efficacy and Safety of Dapoxetine in the Treatment of Subjects With Premature Ejaculation — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=572&filename=CR004231_CSR.pdf